CLINICAL TRIAL: NCT03615521
Title: Diz Osteoartritinde Farklı Proprioseptif Nöromüsküler Fasilitasyon Tekniklerinin, Ağrı, Propriosepsiyon, Postural Kontrol, Kas Kuvveti, Eklem Hareket Açıklığı ve Diz Fonksiyonları Üzerine Olan Etkileri
Brief Title: Different Proprioceptive Neuromuscular Facilitation (PNF) Technique in Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karamanoğlu Mehmetbey University (Other)
Responsible Party: Principal Investigator, Ayşenur Gökşen, Research Assistant, Karamanoğlu Mehmetbey University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2017/09-36 (KA-17112)
Record Dates: First submitted 2017-12-11; First posted 2018-08-06 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-02

CONDITIONS: Muscle Weakness; Balance Disorders; Knee Pain; Knee Osteoarthritis
MeSH Terms: conditions — Muscle Weakness; Osteoarthritis, Knee | interventions — High-Energy Shock Waves

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Repeated Contraction Exercise Group (Experimental): Repeated Contractions Exercise Group, Hotpack apply for knee 20 minute, Ultrasound is a termal ajan which use for 10 minute and Repeated Stretch (Repeated Contractions) exercise. Repeated Contractions exercise is type of Proprioceptive Neuromusculer Facilititation Exercise. 3 session for 6 weeks.
  Interventions: Other: Hotpack; Other: Ultrasound; Other: Repeated Contraction Exercise
- Combine Exercise Group (Experimental): Combination of Isotonics Exercise Group, Hotpack apply for knee 20 minute, Ultrasound is a termal ajan which use for 10 minute Combination of Isotonics Exercise. Combination of Isotonics Exercise is type of PNF. Combined concentric, eccentric, and stabilizing contractions of one group of muscles (agonists) without relaxation.
  3 Session for 6 weeks.
  Interventions: Other: Hotpack; Other: Ultrasound; Other: Combine Exercise
- Standart Exercise Therapy (Experimental): Classic Physiotherapy: Hotpack, Ultrasound, Standart exercise program to improve Quadriceps, Hamstring and hip muscle strength.
  3 session for 6 weeks.
  Interventions: Other: Hotpack; Other: Ultrasound; Other: Standart Exercise Therapy

INTERVENTIONS:
Other: Hotpack — Hotpack applied 20 minutes for knee 3 session for 6 weeks
Other: Ultrasound — Ultrasound applied 10 minutes for knee 3 session for 6 weeks
Other: Combine Exercise — Proprioceptive Neuromusculer Facilitation Technique İnclude eccentric and concentric contractions 3 session for 6 week
  Arms: Combine Exercise Group
Other: Repeated Contraction Exercise — Proprioceptive Neuromusculer Facilitation Technique include concentric contractions 3 session for 6 week
  Arms: Repeated Contraction Exercise Group
Other: Standart Exercise Therapy — Quadriceps, hamstring and hip muscle strength exercise. Hamstring stretch exercise.
  3 session for 6 week
  Arms: Standart Exercise Therapy

SUMMARY:
The aim of this study is to investigate the effects of 6-week physiotherapy and rehabilitation programs involving different 'Proprioceptive Neuromuscular Facilitation' (PNF) techniques in patients with knee osteoarthritis on pain, proprioception, postural control, muscle strength, range of motion and knee functions

DETAILED DESCRIPTION:
The results obtained from this study will contribute to the selection of PNF technique which is most suitable for physiotherapies working on knee osteoarthritis in clinics as well as demonstrating the efficacy of PNF which has been studied in the literature very few times.

As a result of this study, the evidence value of the PNF technique will be determined in the physiotherapy and rehabilitation program of patients with knee osteoarthritis, and the efficacy of this technique, which is theoretically adopted, will be demonstrated scientifically. It will also determine the most ideal of the two PNF techniques to be applied in patients with knee osteoarthritis

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 45-65
* The diagnosis of stage 1-2 osteoarthritis by the orthopedist
* Volunteerig for research
* No hearing, vision and speech impediment

Exclusion Criteria:

* Patients with intra-articular contracture,
* No Meniscus and no ligament problems
* Presence of any neurological or cardiopulmonary disease that may affect the results of the study

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-01-20 (Actual); Primary Completion 2021-05-20 (Actual); Study Completion 2021-11-10 (Actual)

PRIMARY OUTCOMES:
Quadriceps Femoris Muscle Strength | 6 week
  Quadriceps Femoris muscle strength is evaluated Biodex System. Patients performs knee extension strongly and system analyzed. System gives us Peak Torque which indicates the muscle's maximum strength capability.
  1 repetition maximum (RM) isotonic strength test.

SECONDARY OUTCOMES:
Knee Proprioception (30-45 and 60 degree) | 6 week
  Proprioception is evaluated with Biodex System (30-45 and 60 degree)
KOOS score | 6 week
  KOOS consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL). The previous week is the time period considered when answering the questions. Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale (scoring instructions are available in a separate document: KOOS Scoring). A total score has not been validated and is not recommended.
Step test | 6 week
  Climb and step in 10 steps. Brief time is better.
Womac Score | 6 week
  It is a self-administered questionnaire consisting of 24 items divided into 3 subscales Pain (5 items): during walking, using stairs, in bed, sitting or lying, and standing upright Stiffness (2 items): after first waking and later in the day Physical Function (17 items): using stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on / taking off socks, rising from bed, lying in bed, getting in / out of bath, sitting, getting on / off toilet, heavy domestic duties, light domestic duties scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function. Usually a sum of the scores for all three subscales gives a total WOMAC score, however there are other methods that have been used to combine scores.
  Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
6 Minute walking test | 6 week
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity. "The object of this test is to walk as far as possible for 6 minutes. More walk in a short time is better performance.
Balance | 6 week
  Balance is evaluated Biodex Balance System (BBS). This device, clinicians can assess neuromuscular control by quantifying the ability to maintain dynamic bilateral and unilateral postural stability on a static or unstable surface. In the measurement with the BBS, the personal values of the patient are determined and compared to reference values. Balance deficits are determined on this basis. BBS permits three measurements to be obtained including overall stability index (OSI), anterior-posterior stability index (APSI) and medial-lateral stability index (MLSI). Balance and risk of fall were assessed using two trials over a period of 30 seconds with 10 seconds rest in between. If total score close zero, accepted better.
Knee Pain Severity | 6 week
  Pain is evaluated with visual analog scale. The pain VAS is self-completed by the respondent. The respondent is asked to place a line perpendicular to the VAS line at the point that represents their pain intensity. ''0'' means no pain, ''10'' means much pain, ''5'' means moderate pain.
Algometer | 6 week
  Algometers are devices that can be used to identify the pressure and/or force eliciting a pressure-pain threshold.The handheld algometer had a 1-cm2 round rubber application surface.The investigator placed the digital pressure algometer on a site to be inspected and pressed against the tester in a vertical direction while increasing the force at a constant rate of 1 kg/cm2. The investigator instructed the subjects to express pain either by saying "ouch" or raising their hands when only slight pain was felt.

OTHER OUTCOMES:
Time up and go test | 6 week
  Patient stand up, walk to the line on the floor and turn around and walk back to the chair and sit down. Start timing on the word "GO" and stop timing when the subject is seated again correctly in the chair with their back resting on the back of the chair.
  Normal healthy elderly usually complete the task in ten seconds or less. Very frail or weak elderly with poor mobility may take 2 minutes or more.

CONTACTS AND LOCATIONS:
Overall Officials: Filiz Can, Prof., Study Director — Hacettepe University
Locations (1):
- Hacettepe, Ankara, Turkey (Türkiye)